CLINICAL TRIAL: NCT01374438
Title: A 3-month Randomized, Double-Blind, Placebo-Controlled, Feasibility Study to Evaluate the Effects of MSDC-0160 on Brain Glucose Utilization, Cognition, Safety and Tolerability in Older Persons With Mild Alzheimer's Disease
Brief Title: 3-month Study of MSDC-0160 Effects on Brain Glucose Utilization, Cognition & Safety in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metabolic Solutions Development Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSDC-0160-C006
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; cognitive function; brain glucose utilization; FDG-PET
MeSH Terms: conditions — Alzheimer Disease | interventions — MSDC-0160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSDC-0160 capsules (Experimental): MSDC tablets contained in #00 capsules
  Interventions: Drug: MSDC-0160
- Placebo capsules (Placebo Comparator): Placebo tablets contained in #00 capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSDC-0160 — MSDC-0160 150 mg capsules given once daily for 90 days
  Other Names: Mitoglitazone
  Arms: MSDC-0160 capsules
Drug: Placebo — Placebo capsules given once daily for 90 days
  Arms: Placebo capsules

SUMMARY:
This study will evaluate the effect of 150 mg MSDC-0160 taken daily for 90 days compared to the effect of placebo on changes in brain glucose utilization using FDG-PET and cognition in older persons with mild Alzheimer's disease. Safety and tolerability of MSDC-0160 in this population will also be studied. These results will be used to design larger studies of MSDC-0160 in persons with mild Alzheimer's disease.

DETAILED DESCRIPTION:
The specific objective is to examine the feasibility of conducting future large scale studies on the efficacy of MSDC-0160 in persons with mild Alzheimer's disease. Efficacy and safety will be assessed as follows:

1. Estimate the effect size of 150 mg daily MSDC-0160 versus placebo on 3-month change in brain glucose utilization using FDG-PET pre-specified regions of interest analysis. The a priori regions of interest (ROI) will include five bilateral regions: posterior cingulate, parietal cortex (angular gyrus), lateral temporal cortex, medial temporal cortex, and anterior cingulate-medial frontal cortex.
2. Estimate the effect size of MSDC-0160 versus placebo on 3-month change in brain glucose utilization, using FDG-PET voxel-based analysis.
3. Estimate the effect size of MSDC-0160 treatment versus placebo on 3-month change in cognitive function as determined by global cognitive function on a neuropsychological battery of 19 tests.
4. Estimate the effect size of MSDC-0160 versus placebo on 3-month change in cognitive function as determined by the ADAS-Cog subscale.
5. Estimate the effect of 3-months of MSDC-0160 treatment versus placebo on a 9-item executive function scale.
6. Explore whether baseline levels of peripheral inflammatory biomarkers (HMW adiponectin, TNFα, IL-6, hsCRP, and FFA) or genotypes including, but not limited to, the apolipoprotein ε4 allele explain the heterogeneity in baseline level of brain glucose utilization and, in MSDC-0160 users, 3-month brain glucose utilization.
7. Explore whether changes in peripheral inflammatory biomarkers correlate with changes in 3-month brain glucose utilization in MSDC-0160 users.
8. Investigate the safety of MSDC-0160 versus placebo using reports of early study termination and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females 55-85 years of age.
2. Females should be either postmenopausal or surgically sterilized. Males with female partners of child-bearing potential must use contraception if engaging in sexual intercourse.
3. Diagnosis of probable Alzheimer's disease based on NIA-AA criteria with MMSE scores of 20 or greater.
4. Willing and able to take part in up to six study visits over a 5-month period, with the support of a caregiver as needed.
5. Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study, with the support of a caregiver as needed.

Exclusion Criteria:

1. Diagnosis of diabetes, including use of anti-diabetic medications, or fasting plasma glucose >125 mg/dl or Hemoglobin A1c>6.4%.
2. Unable to participate in FDG-PET scanning, including:

   * Inability to cooperate/claustrophobia (no sedation offered for this protocol).
   * Inability to lie still on the scanner bed for 40 minutes.
   * Total radiation dose exposure to the subject in any given year exceeds the limits of annual and total dose commitment of 50 mSv (5 REMs). The two FDG-PET scans will result in an approximate exposure of 10 mSv (1 REM).
3. Diagnosis of significant neurological/psychiatric disease other than AD, including, but not limited to, any of the following: vascular dementia according to NINDS-AIREN criteria, space occupying cerebral lesion, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, and seizures.
4. History of heart failure (including CHF).
5. Previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 6 months prior to screening.
6. Inability to undergo a clinical (1.5T) MRI of the brain without contrast and lack of a usable (less the 12 months prior to screening) MRI on record. Contraindications to undergoing an MRI of the brain include, but are not limited to, pacemakers; implantable cardioverter defibrillators; cochlear implants; cerebral aneurysm clips; implanted infusion pumps; implanted nerve stimulators; metallic splinters in the eye; and, other magnetic, electronic or mechanical implants or clinical findings that in the judgment of the investigator would pose a potential hazard in combination with MRI.
7. ALT and/or AST levels that are twice the upper limit of normal; bilirubin levels that exceed 2 mg/dL; serum creatinine >1.5 mg/dL in men or > 1.4 mg/dL in women.
8. Current or history of severe or unstable disorder (medical or psychiatric) requiring treatment that may make the subject unlikely to complete the study.
9. Malignancy (other than non-melanoma skin cancer) within the last 5 years.
10. Known history of HIV, hepatitis B, or hepatitis C.
11. Blood pressure greater than 160/100 mmHg. Subjects with elevated BP will be allowed at the discretion of the principal investigator. Individuals with hypertension must have been stabilized to the current treatment regimen for at least 6 weeks prior to screening and not need adjustments to their treatment regimen during the entire study period.
12. Change in other medications to treat Alzheimer's disease within 3 months prior to screening. Change in medication to treat other conditions within 6 weeks prior to screening or during the study period.
13. Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds, or any of their stated ingredients.
14. History of alcohol or drug abuse within 6 months of screening.
15. Have participated in an investigational study or received an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
16. Single 12-lead ECG demonstrating a QTcB >450 msec or other clinically significant finding at screening. A single repeat ECG may be done at the investigator's discretion.
17. Any surgical or medical condition which may significantly alter the absorption of any drug substance including, but not limited to, any of the following: history of major gastrointestinal tract surgery, currently active inflammatory bowel syndrome.
18. Evidence of clinically relevant pathology that in the investigator's opinion could interfere with the study results or put the subject's safety at risk.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Colca, PhD, Study Director — MSDC; Raj C. Shah, MD, Principal Investigator — Rush Memorial University Medical Center
Locations (1):
- Rush Memorial University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Shah RC, Matthews DC, Andrews RD, Capuano AW, Fleischman DA, VanderLugt JT, Colca JR. An evaluation of MSDC-0160, a prototype mTOT modulating insulin sensitizer, in patients with mild Alzheimer's disease. Curr Alzheimer Res. 2014;11(6):564-73. doi: 10.2174/1567205011666140616113406. PMID 24931567

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Started | 16 | 13
Completed | 16 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects completed the full study and are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | MSDC-0160 Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (8.8) | 71.0 (8.0) | 71.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Presence of an Apolipoprotein E e4 allele [Number; unit: participants]
  Apo E e4 allele present | 10 | 9 | 19
  Apo E e4 allelle absent | 6 | 4 | 10
Mini-Mental State Examination Score [Mean (Standard Deviation); unit: units on a scale] — Screening Mini-Mental State Examination Score, Mean (SD). Possible scores range between 0 and 30. Scores ≥27 indicate normal cognition, 19-24 indicate mild impairment, 10-18 indicate moderate impairment, and scores ≤9 indicate severe impairment.
  units on a scale | 22.8 (2.4) | 25.2 (2.1) | 23.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Effects of MSDC-0160 on Cerebral Metabolic Glucose Rate or Placebo Over 12 Weeks in Pre-specified Regions of Interest Analysis Referenced to Cerebellum
Description: Investigate the effect of 150 mg daily MSDC-0160 vs placebo on 3-month change in brain glucose utilization using FDG-PET pre-specified regions of interest analysis referenced to cerebellum, including five bilateral regions: posterior cingulate, parietal cortex (angular gyrus), lateral temporal cortex, medial temporal cortex, and anterior cingulate-medial frontal cortex. Results are reported as Standardized Uptake Value Ratios. A change from baseline in the metabolic rate of glucose that is ≥0 indicates maintenance of brain glucose utilization, whereas values <0 indicate a decline in brain glucose utilization.
Time Frame: Days 1(baseline) and 91
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Number analyzed (Participants) | 16 | 13
Ratio
  Posterior cingulate | 0.01 (0.03) | -0.02 (0.03)
  Parietal cingulate | 0.01 (0.02) | -0.03 (0.03)
  Lateral temporal cortex | 0.00 (0.02) | -0.02 (0.03)
  Medial temporal cortex | 0.01 (0.02) | -0.01 (0.02)
  Ant. cing.-frontal cortex | 0.00 (0.02) | -0.03 (0.03)

2. Secondary Outcome: Change From Baseline in Global Cognitive Function Tests
Description: Change from baseline in cognitive function, as determined by global cognitive function on a neuropsychological battery of 19 tests, following 3 months treatment with MSDC-0160 versus placebo. A summary measure of global cognitive function was constructed by converting raw scores from 19 individual tests into z-scores as described by Bennett DA, et al., The Rush Memory and Aging Project: study design and baseline characteristics of the study cohort, Neuroepidemiology. 2005;25(4):163-175.
Time Frame: Days 1 (baseline) and 91
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Number analyzed (Participants) | 16 | 13
z-scores | -0.06 (0.11) | 0.03 (0.59)

3. Secondary Outcome: Change From Baseline in Cognitive Function as Determined by the ADAS-Cog Subscale
Description: Alzheimer's Disease Assessment Scale - Cognitive Subscale, an assessment of cognitive ability. Scores on 11 individual tasks were summed to produce the reported total score, with a possible range of 0 (no impairment) to 70 (severe impairment).
Time Frame: Days 1 (baseline) and 91
Population: One subject in the MSDC-0160 group and 2 subjects in the placebo group were not able to complete the ADAS-Cog tests at both study time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Number analyzed (Participants) | 15 | 11
Scores on a scale | 0.69 (3.62) | 2.21 (2.87)

4. Secondary Outcome: Change From Baseline in Cognitive Function as Estimate With the Executive Function Scale
Description: Estimate of the effect of 3-months of MSDC-0160 treatment versus placebo on a 9-item executive function scale. A summary measure of executive function was constructed by converting raw scores from 9 individual tests into z-scores as described by Bennett DA, et al., The Rush Memory and Aging Project: study design and baseline characteristics of the study cohort, Neuroepidemiology. 2005;25(4):163-175.
Time Frame: Days 1 (baseline) and 91
Population: One subject in the MSDC-0160 group and 2 subjects in the placebo group were not able to complete the executive function tests at both study time points.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Number analyzed (Participants) | 15 | 11
z-score | -0.04 (0.25) | 0.00 (0.45)

5. Secondary Outcome: Change From Baseline in HMW Adiponectin of MSDC-0160 or Placebo Over 12 Weeks
Description: Estimate the effect of 150 mg daily MSDC-0160 versus placebo on levels of high molecular weight adiponectin. Increases in HMW adiponectin suggest improved insulin sensitivity.
Time Frame: Days 1(baseline) and 91
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Number analyzed (Participants) | 16 | 13
micromol/L | 17822 (10940) | 795 (4477)

ADVERSE EVENTS:
Time Frame: Collection of safety data began in August 2011, when the first subject was randomized, and continued until March 19, 2013, when all 29 subjects had completed all study activities.
Description: Subjects were asked to report any adverse events during each study visit.
Arm/Group | MSDC-0160 Capsules | Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/13
Other Adverse Events (participants affected / at risk) | 7/16 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSDC-0160 Capsules (N=16) | Placebo Capsules (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSDC-0160 Capsules (N=16) | Placebo Capsules (N=13)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Peripheral Edema (General disorders) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoechoic nodule (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Scrotal varicose vein rupture (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Patent foramen ovale (Cardiac disorders) | 0 (0) | 1 (1)
QTcB elevation (Cardiac disorders) | 0 (0) | 1 (1)
Cognitive decline, subjective (Nervous system disorders) | 0 (0) | 1 (1)
Syncope, vasovagal (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less